CLINICAL TRIAL: NCT01124591
Title: Clinical Trial to Determine the Effect of a Brief Behavioral Intervention in Reducing Drug Misuse Among an Emergency Department Population
Brief Title: Brief Intervention for Drug Misuse in the Emergency Department
Acronym: BIDMED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roland C. Merchant, MD. MPH, ScD, Attending Physician, Rhode Island Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 0113-09
Record Dates: First submitted 2010-05-10; First posted 2010-05-17 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Substance Abuse Detection; HIV; Hepatitis B; Hepatitis C; Brief Intervention; HIV Infections
MeSH Terms: conditions — Hepatitis B; Hepatitis C; HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Assessment and brief intervention
  Interventions: Behavioral: Brief motivational intervention

INTERVENTIONS:
Behavioral: Brief motivational intervention — two session delivered two weeks apart

SUMMARY:
Although screening, brief intervention, and referral to treatment (SBIRT) approaches are effective in reducing alcohol misuse and its associated risk-taking behaviors and negative consequences, there is little research demonstrating the effectiveness of SBIRT for illicit and/or prescription drug misuse. Misusers of illicit and/or prescription drugs frequently seek medical care in emergency departments (EDs), particularly for reasons related to their misuse. As a result, the ED is well suited as a site to conduct an analysis of the effectiveness of SBIRT for this population.

The Brief Intervention for Drug Misuse for the Emergency Department (BIDMED) study is a randomized, controlled, trial that will include adult ED patients at a large, academic, trauma center (Rhode Island Hospital) and a community hospital (The Miriam Hospital) who have a subcritical illness or injury and whose screening indicates illicit and/or prescription drug misuse. BIDMED participants will be randomized to receive screening only (SO) or brief intervention (BI) with appropriate referral to treatment. Participants will complete a battery of blinded baseline assessments using standardized instruments as well as adapted instruments specific to the aims of this study. All participants will undergo blinded follow-up assessments at three, six, and twelve months post-randomization. The primary hypotheses addressed in the BIDMED study are that, compared to participants in the SO arm, participants in the BI arm will show a significantly greater reduction in: (1) drug misuse within the prior 30 days at three months post-randomization, (2) behaviors associated with drug misuse at six months post-randomization; and (3) negative physical health, psychosocial health, and socioeconomic consequences at twelve months post-randomization. As a secondary aim, the impact of BI compared to SO will be assessed on participants contacting, enrolling in, and completing a drug treatment program. In addition, the impact of BI compared to SO on increasing uptake of HIV and hepatitis B/C screening will be measured. A mechanisms of change model that addresses the expected mediators and moderators of change to explain the effects of SBIRT in this setting will also be developed and tested. Further, the epidemiology of illicit and/or prescription drug misuse will be assessed in a random sample of ED patients.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of illicit and/or prescription drug misuse in the past three-months. Presenting at the emergency department for medical care.

Exclusion Criteria:

Not age appropriate, in custody, medically unstable, actively psychotic, suicidal

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1030 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in past 30 day drug misuse | 12 months post-randomization
Reduction in behaviors associated with drug misuse | 12 months post-randomization
Reduction negative physical health, psychosocial health, and socioeconomic consequences | 12 months post-randomization

SECONDARY OUTCOMES:
Uptake of HIV and hepatitis B/C screening | 3 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD; ScD, Principal Investigator — Rhode Island Hospital; Ted Nirenberg, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Merchant RC, Zhang Z, Zhang Z, Liu T, Baird JR. Lack of efficacy in a randomised trial of a brief intervention to reduce drug use and increase drug treatment services utilisation among adult emergency department patients over a 12-month period. Emerg Med J. 2018 May;35(5):282-288. doi: 10.1136/emermed-2016-206540. Epub 2018 Feb 2. PMID 29437758
- [Derived] Guan W, Liu T, Baird JR, Merchant RC. Evaluation of a brief intervention to reduce the negative consequences of drug misuse among adult emergency department patients. Drug Alcohol Depend. 2015 Dec 1;157:44-53. doi: 10.1016/j.drugalcdep.2015.10.007. Epub 2015 Oct 13. PMID 26482090
- [Derived] Merchant RC, Baird JR, Liu T. Short-term Efficacy of a Brief Intervention to Reduce Drug Misuse and Increase Drug Treatment Utilization Among Adult Emergency Department Patients. Acad Emerg Med. 2015 Oct;22(10):1172-80. doi: 10.1111/acem.12767. Epub 2015 Sep 16. PMID 26375468
- [Derived] Bernardino VL, Baird JR, Liu T, Merchant RC. Comparison of substance-use prevalence among Rhode Island and The Miriam Hospital Emergency Department patients to state and national general population prevalence estimates. R I Med J (2013). 2014 Apr 1;98(4):30-4. PMID 25830171
- [Derived] Merchant RC, Baird JR, Liu T, Taylor LE. HCV among The Miriam Hospital and Rhode Island Hospital Adult ED Patients. R I Med J (2013). 2014 Jul 1;97(7):35-9. PMID 24983020